CLINICAL TRIAL: NCT06312930
Title: Neuromodulation of Transcranial Pulse Stimulation on Primary Motor Cortex in Adults: A Randomized, Cross-over, Single-blind, Sham-controlled, Pilot Trial
Brief Title: Transcranial Pulse Stimulation on Motor Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20220816001-03
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-12

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real TPS group (Experimental): 1. Healthy adults aged 18-65 years old will receive one single session of real TPS on the primary motor cortex.
  2. Before and after TPS, participants will perform two visuomotor tasks (a simple reaction time task and a nine-hole peg test).
  3. The stimulation target on the primary motor cortex will be determined by transcranial magnetic stimulation (TMS). Measurements of the resting motor threshold by TMS will be conducted for each participant before the real TPS session.
  Interventions: Device: Transcranial pulse stimulation
- Sham TPS group (Sham Comparator): Sham stimulation comprises TPS on the vertex as the control region (sham control).
  Stimulation duration, intensity, as well as pre- and post stimulation assessments are the same as in the experimental arm.
  In this cross-over study, the order of the real and sham stimulation conditions will be randomized and separated by 24 hours.
  Interventions: Device: Transcranial pulse stimulation

INTERVENTIONS:
Device: Transcranial pulse stimulation — A single session of TPS will be performed, applying 1000 pulses in the session (single ultrashort (3 μs) ultrasound pulses, 0.2-0.25 mJ mm-2, ~5 Hz pulse frequency)

SUMMARY:
Transcranial pulse stimulation (TPS) is a newly developed non-invasive brain stimulation (NIBS) technique from Austria & Germany with highly promising applicability in neuropsychiatric disorders. Clinical trials have shown a beneficial effect of TPS in patients with Alzheimer's disease and depression. However, the mechanism of action of TPS treatment is unknown. There is a lack of controlled studies with sufficient sample size to draw reliable conclusions on the modulatory effect of TPS. The primary motor cortex is a common target when investigating the neuromodulation effect of NIBS techniques. Here, a randomized, cross-over, single-blind, sham-controlled clinical trial is proposed to probe the effects of TPS over the primary motor cortex on modulating motor response and motor behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* No physical, neurological or psychiatric disorder
* Right-handedness

Exclusion Criteria:

* Background with neuroscience
* TPS and TMS contraindications, including metal implants, pregnancy, coagulation disorders, thrombosis, brain tumor, cortisone therapy up to 6 weeks before first stimulation, pacemakers or cochlear implants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Change in movement time in nine-hole peg test after TPS | Immediately after the completion of the single session TPS, 10 minutes after the single session TPS, 20 minutes after the single session TPS, 30 minutes after the single session TPS, 40 minutes after the single session TPS
  Primary clinical outcome measure will be a change in movement time in nine-hole peg test after TPS. Less movement time is indicative of greater improvement in hand dexterity and motor function.
Change in reaction time in Deary-Liewald reaction time task after TPS | Immediately after the completion of the single session TPS, 10 minutes after the single session TPS, 20 minutes after the single session TPS, 30 minutes after the single session TPS, 40 minutes after the single session TPS
  Primary clinical outcome measure will be a change in reaction time in Deary-Liewald reaction time task after TPS. Less reaction time is indicative of greater improvement in motor function.

SECONDARY OUTCOMES:
The influence of motor excitability measured by resting motor threshold (RMT) on post-TPS motor performance | 30 minutes before TPS session, immediately after the completion of the single session TPS, 10 minutes after the single session TPS, 20 minutes after the single session TPS, 30 minutes after the single session TPS, 40 minutes after the single session TPS
  The RMT will be measured before the TPS, which is indicative of the motor excitability. The investigators will explore the correlation between the RMT and post-TPS motor performance measured by the nine-hole peg test; as well as explore correlation between RMT and post-TPS motor performance measured by the Deary-Liewald reaction time task.

CONTACTS AND LOCATIONS:
Overall Officials: Georg S. Kranz, PhD, Principal Investigator — The Polytechnic University
Locations (1):
- Georg Kranz, PhD, Hong Kong, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin PP, Chak IK, Kan RL, Jin MX, Zhang BB, Xia AW, Lin TT, Wang SX, Liu JH, Cheung T, Kranz GS. Effects of Transcranial Pulse Stimulation of the Primary Motor Cortex on Motor Performance in Healthy Adults: A Randomized Crossover Pilot Study. CNS Neurosci Ther. 2025 Dec;31(12):e70711. doi: 10.1002/cns.70711. PMID 41420421